CLINICAL TRIAL: NCT03261245
Title: Hypertension Disorders During Pregnancy and Multi-exposure to Environmental Noise and Atmospheric Pollution in an Urban Setting: Case-control Study in Women Who Gave Birth at Dijon and Besançon CHUs Between 2005 and 2009
Brief Title: Relationship Between Multi-exposure to Noise and Air Pollution and the Onset of Hypertension Disorders During Pregnancy
Acronym: HTA-BQuA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MARIET AOI 2016
Record Dates: First submitted 2017-08-23; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Women Who Gave Birth at Dijon and Besançon CHUs Between 2005 and 2009

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cas: Onset of a hypertension disorder during pregnancy
- Controls: No hypertension disorder during pregnancy

SUMMARY:
This retrospective study aimed to analyse the relationship between multi-exposure to noise and air pollution the onset of hypertension disorders during pregnancy

It will be conducted in 2650 mothers who gave birth at Dijon or Besançon CHU between 2005 and 2009 split into two groups:

* 530 cases (women who experienced hypertension disorders during pregnancy
* 2120 controls (women who did not experience a hypertension disorder during pregnancy)

ELIGIBILITY:
Inclusion Criteria:

* Women living in Besançon or one of the 15 communes of the Dijon conurbation
* Who gave birth at Dijon or Besançon CHU
* Between 1st January 2005 and 31st December 2009

Criterion for the inclusion of cases:

* Onset of a hypertension disorder during pregnancy defined according to expert recommendations

Criterion for the inclusion of controls:

* No hypertension disorder during pregnancy

Exclusion Criteria:

* Medical termination of pregnancy
* Opposition to the use of their data

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women who gave birth at Dijon and Besançon CHU between 2005 and 2009
Sampling Method: Non-Probability Sample
Enrollment: 2650 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Onset of a hypertension disorder during pregnancy | at baseline

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de BESANCON, Besançon
  - CHU Dijon Bourgogne, Dijon